CLINICAL TRIAL: NCT02711436
Title: Fast Magnetic Resonance Imaging as Compared to Computed Tomography Scan in Pediatric Orbital Cellulitis Imaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HYMC-0022-16
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Orbital Cellulitis
MeSH Terms: conditions — Orbital Cellulitis | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computed Tomography Scan (Active Comparator): To determine the presence of periosteal or orbital abscess, intracranial abscess and dural venous sinus thrombosis that are imaged properly with Computed Tomography scan.
  Interventions: Device: Computed Tomography Scan
- Fast Magnetic Resonance Imaging (Active Comparator): To determine the presence of periosteal or orbital abscess, intracranial abscess and dural venous sinus thrombosis that are imaged properly with T1/T2-weighted MRI.
  Interventions: Device: Fast Magnetic Resonance Imaging

INTERVENTIONS:
Device: Computed Tomography Scan
  Arms: Computed Tomography Scan
Device: Fast Magnetic Resonance Imaging
  Arms: Fast Magnetic Resonance Imaging

SUMMARY:
The aim of the study is to compare orbital and central nervous system (CNS) imaging with Computed Tomography (CT) scan to that of Fast Magnetic Resonance Imaging (Fast MRI) in children with mild, moderate or severe orbital cellulitis with medical indications for imaging.

ELIGIBILITY:
Inclusion Criteria:

* Children with orbital cellulitis with indications for imaging

Exclusion Criteria:

* All others

Ages: 6 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
MRI sensitivity for the detection of orbital cellulitis compared to CT | One year
  MRI results will be compared to CT results

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Cohen, MD, PhD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No